CLINICAL TRIAL: NCT00154297
Title: A National Multicentre Randomized Study Comparing the Early Versus Delayed Administration of Everolimus in de Novo Kidney Transplant Recipients at Risk of Delayed Graft Function
Brief Title: Efficacy and Safety of Early Versus Delayed Administration of Everolimus in de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2420
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-03

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation; everolimus; immunosuppressants; wound-healing
MeSH Terms: interventions — Everolimus

ARMS (2):
- Immediate Everolimus (Active Comparator): Patients received Everolimus starting within 48 hours of kidney transplant through to the end of the study, administered orally twice a day. Dose was adjusted in order to maintain a trough level between 3-8 ng/mL.
  Interventions: Drug: Everolimus (RAD001)
- Delayed Everolimus (Experimental): Patients received Everolimus 4 weeks after kidney transplant until the end of the study, administered orally twice a day. The dose was adjusted in order to maintain a trough level between 3-8 ng/mL. Patients received mycophenolic acid until everolimus was initiated.
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001)

SUMMARY:
The purpose of this study is to evaluate if the delayed administration of everolimus could reduce the everolimus associated "anti-proliferative complications" (e.g. wound healing disorder) while maintaining efficacy, when compared to the immediate administration of everolimus in de novo renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of cadaveric kidney transplants
* Patients at risk of DGF defined as one or more of the following:

  * Donor age > 55 years
  * Cold ischemic time (CIT) ≥ 24 hours but < 40 hours
  * Second or subsequent renal transplantation

Exclusion Criteria:

* Patients who have received an investigational drug within 4 weeks of baseline period
* Patients who are recipients of multiple organ transplants, including more than one kidney, or previous transplant with any organ other than kidney
* Patients with body mass index (BMI) > 32 kg/m2

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Everolimus | Delayed Everolimus
Started | 65 (Randomized population.) | 74 (Randomized population.)
Completed | 57 (Completed study by 12 month.) | 67 (Completed study by 12 month.)
Not Completed | 8 | 7
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Everolimus | Delayed Everolimus | Total
Number analyzed (Participants) | 65 | 74 | 139
Age Continuous [Mean (Standard Deviation); unit: years] — baseline measure based on randomized population.
  years | 57.3 (10.46) | 58.4 (9.86) | 57.9 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measure based on randomized population.
  Participants
    Female | 19 | 20 | 39
    Male | 46 | 54 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Considered in Failure for the Primary Failure Endpoint at 3 Months
Description: "In Failure", is at least one of these events occurred within the first 3 months: delayed graft function(DGF), (need for dialysis within the first 7 days,minus day one,post-transplantation); Biopsy proven acute rejection (BPAR), Graft loss, (allograft was presumed lost on the day the patient started and not removable from dialysis). Death; Loss to follow-up; Wound healing disorder(Any wound related to the kidney transplantation being opened beyond 3 weeks, or infected, or drained fluid or herniated was considered not healed).
Time Frame: Month 3
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 65 | 74
Participants
  Failure at month 3 - Total | 36 | 47
  Dialysis within first 7 days | 16 | 18
  Efficacy failure (Total) | 14 | 15
  --BPAR | 7 | 7
  --Graft Loss | 5 | 3
  --Death | 4 | 2
  --Lost to follow-up (composite efficacy endpoint) | 0 | 4
  Wound healing disorder | 24 | 28
  Loss to follow-up for the primary failure endpoint | 0 | 3

2. Secondary Outcome: Number of Participants Considered in Failure for the Primary Failure Endpoint at 6 Months Post-transplantation.
Description: The primary efficacy variable was the "primary failure endpoint" at 6 months defined as the occurrence of one or more of the following events within the first 6 months:
  * delayed graft function (DGF), defined as the need for dialysis within the first 7 days post-transplantation excluding the first day post-transplantation
  * efficacy failure (biopsy proven acute rejection (BPAR), graft loss, death or loss to follow-up)
  * wound healing disorder related to initial transplant surgery
Time Frame: at 6 Month post-transplantation
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 65 | 74
Participants
  Failure at month 6 - Total | 39 | 48
  Dialysis within first 7 days | 16 | 18
  Efficacy failure (Total) | 17 | 22
  --BPAR | 10 | 13
  --Graft Loss | 5 | 4
  --Death | 4 | 2
  --Lost to follow-up (composite efficacy endpoint) | 0 | 4
  Wound healing disorder | 25 | 28
  Loss to follow-up for the primary failure endpoint | 0 | 3

3. Secondary Outcome: Number of Participants Considered in Failure for the Primary Failure Endpoint at 12 Months Post-transplantation.
Description: The primary efficacy variable was the "primary failure endpoint" at 12 months defined as the occurrence of one or more of the following events within the first 12 months:
  * delayed graft function (DGF), defined as the need for dialysis within the first 7 days post-transplantation excluding the first day post-transplantation
  * efficacy failure (biopsy proven acute rejection (BPAR), graft loss, death or loss to follow-up)
  * wound healing disorder related to initial transplant surgery
Time Frame: at 12 Month post-transplantation
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 65 | 74
Participants
  Failure at month 12 - Total | 42 | 49
  Dialysis within first 7 days | 16 | 18
  Efficacy failure (Total) | 22 | 25
  --BPAR | 13 | 15
  --Graft Loss | 6 | 5
  --Death | 5 | 2
  --Lost to follow-up (composite efficacy endpoint) | 0 | 5
  Wound healing disorder | 26 | 28
  Loss to follow-up for the primary failure endpoint | 0 | 3

4. Secondary Outcome: Number of Participants Who Underwent Any Dialysis Within the 12-month Treatment Period
Description: The number of patients who underwent any dialysis within the 12-month treatment period.
Time Frame: Month 12
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 65 | 74
Participants | 16 | 24

5. Secondary Outcome: Duration of Dialysis
Description: The mean duration in days of any dialysis session that occurred within the 12 month treatment period.
Time Frame: 12 months
Population: The number of patients analyzed includes those with any dialysis in the 12 month period
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 16 | 24
Days | 11.9 (7.01) | 7.8 (7.42)

6. Secondary Outcome: Number of Participants With Any Wound Healing Disorder During the 12-month Treatment Period
Description: A wound was considered healed if all the suture material and staples were removed and the wound was intact by 3 weeks. Any wound opened beyond this point, infected, drained fluid or herniated was considered not healed.
Time Frame: Month 12
Population: Intention to treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Immediate Everolimus | Delayed Everolimus
Number analyzed (Participants) | 65 | 74
Participants
  Any wound healing disorder -Total | 28 | 32
  Wound healing disorder related to transplant | 26 | 28
  Wound healing disorder unrelated to transplant | 2 | 6

ADVERSE EVENTS:
Time Frame: Month 12
Arm/Group | Immediate Everolimus | Delayed Everolimus
Serious Adverse Events (participants affected / at risk) | 45/65 | 57/74
Other Adverse Events (participants affected / at risk) | 64/65 | 70/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Everolimus (N=65) | Delayed Everolimus (N=74)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Retinal artery thrombosis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Implant site haematoma (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 5
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 3 | 6
Abscess (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 1 | 1
Cerebral aspergillosis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 2
Encephalitic infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Genital infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 2 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 2
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Prostate infection (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 6 | 1
Pyelonephritis acute (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 1 | 5
Septic shock (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 5 | 7
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 5 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft loss (Injury, poisoning and procedural complications) | 2 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 6 | 5
C-reactive protein increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 1
Extravasation of urine (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2
Pyelocaliectasis (Renal and urinary disorders) | 1 | 1
Renal aneurysm (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 7
Renal impairment (Renal and urinary disorders) | 4 | 3
Renal tubular disorder (Renal and urinary disorders) | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 2 | 2
Ureteric stenosis (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 4
Lymphocele (Vascular disorders) | 4 | 3
Phlebitis (Vascular disorders) | 1 | 4
Superior vena caval stenosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Everolimus (N=65) | Delayed Everolimus (N=74)
Anaemia (Blood and lymphatic system disorders) | 28 | 33
Leukopenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 12 | 14
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 5 | 4
Oedema peripheral (General disorders) | 26 | 41
Pyrexia (General disorders) | 4 | 1
Bronchitis (Infections and infestations) | 4 | 3
Cytomegalovirus infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 22 | 25
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 15 | 19
Acidosis (Metabolism and nutrition disorders) | 5 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 12 | 15
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 4
Tremor (Nervous system disorders) | 5 | 8
Anxiety (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 3 | 6
Bladder spasm (Renal and urinary disorders) | 1 | 4
Haematuria (Renal and urinary disorders) | 2 | 6
Proteinuria (Renal and urinary disorders) | 8 | 5
Renal impairment (Renal and urinary disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haematoma (Vascular disorders) | 6 | 11
Hypertension (Vascular disorders) | 15 | 17
Lymphocele (Vascular disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.